CLINICAL TRIAL: NCT06639919
Title: Investigation of Biochemical Changes in Maternal Blood as Well as Histological Changes in the Placenta and Amniotic Membrane of Pregnant Women Diagnosed With Preterm Premature Rupture of Membrane
Brief Title: Biochemical and Histological Changes in Pregnant Women With Preterm Premature Rupture of Membrane
Status: Recruiting | Type: Observational
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Other Study IDs: MCBU-PPROM
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Preterm Premature Rupture of Membrane; Placenta Diseases
Keywords: Preterm Premature Membrane Rupture; Premature membrane rupture; Syndecan; Placenta; Amniotic membrane; Proteoglycan
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes; Placenta Diseases; Fetal Membranes, Premature Rupture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Months
Biospecimen Retention: Samples With DNA — placenta tissues and amniotic membrane tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1:: Pregnant women with PPROM
- Group 2:: Control group pregnant women

SUMMARY:
Although preterm premature rupture of membranes (PPROM) is one of the most common causes of preterm birth, it can also lead to serious maternal and neonatal complications. Although there are many known risk factors, the cause is not fully understood . Proteoglycans (PG) are macromolecules containing a core protein and at least one negatively charged polysaccharide glycosaminoglycan side chain and are expressed at high levels in the placenta . Heparan sulfate proteoglycans (HSPG) represent a specific type of PG observed in the placenta. Syndecans (SDC) are the main type of HSPG found in the placenta . There are four types of syndecan, a cell transmembrane PG (syndecan-1, syndecan-2, syndecan-3, syndecan-4) . By containing heparan sulfate and chondroitin sulfate chains, syndecans interact specifically with a variety of ligands, including vascular endothelial growth factor (VEGF), transforming growth factor-beta (TGF-β), and fibronectin, all of which have important functions in the placenta . They play a role in very important physiological processes, including cell proliferation, migration angiogenesis, coagulation system and inflammation .

The aim of this study is to biochemically and histologically investigate the relationship between maternal blood syndecan levels and PPROM, and the relationship between postnatal syndecan levels in the amniotic membrane and placenta and PPROM.

According to our literature review, although there are studies on the presence of syndecan in the amnion and chorion and negative pregnancy outcomes, there are no maternal syndecan blood levels or histopathological examinations regarding PPROM. For this reason, we predict that our study may pave the way for future studies aimed at preventing PPROM and its complications that may occur directly or indirectly. We also think that it will be a pioneer for future studies.

This prospective observational study was conducted by Manisa Celal Bayar University, Department of Gynecology and Obstetrics. The research will be conducted on pregnant women who voluntarily accept to participate in the study.

Group 1: Pregnant women with PPROM (n: 14) Group 2: Control group pregnant women (n: 22) When the planned number of patients is reached, sample collection will be terminated and biochemical and histological examinations will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnancy under 37 weeks
* Age range 18-50
* Being literate in Turkish
* Not having any additional disease
* Agreeing to participate in the study

Exclusion Criteria:

* High-risk pregnancies (gestational hypertension, preeclampsia, HELLP syndrome, chronic hypertension, gestational and pregestational diabetes, cholestasis, intrauterine growth retardation, etc.)
* Multiple pregnancy
* Pregnant women under the age of 18
* Smoking
* Medication use (excluding routinely used food supplements during pregnancy)
* Additional disease (thyroid, renal failure, liver failure, hepatitis, heart disease, connective tissue disease, etc.)
* Immunosuppressive use
* Presence of active or chronic infection
* Presence of active or chronic inflammatory disease
* Patients who gave birth at an external center or later chose to withdraw from the study
* Patients who did not have any exclusion criteria at the time of PPROM or when blood was drawn for the control group, but who later developed any exclusion criteria.
* Premature birth of patients included in the control group

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant Women With Preterm Premature Rupture of Membrane
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
2% women's with PPROM placenta tissues and amnion membrane while birth. Placenta tissues and amnion membrane Staining will be Measured by syndecan 1, 2, 3, 4 immunohistochemistry. | Baseline
maternal and cord blood will be measured by syndecan 1, 2, 3, 4 biochemistry technique. | Baseline

SECONDARY OUTCOMES:
Sociodemographic questions were measured by survey technique. | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Manisa Celal Bayar University, Yunusemre, Mani̇sa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes